CLINICAL TRIAL: NCT03189186
Title: Followed by Nephron-Sparing Surgery or Cytoreductive Nephrectomy in Locally Advanced and Metastatic Renal Cell Carcinomas
Brief Title: Phase-I Trial of Pembrolizumab and Percutaneous Cryoablation Combination Followed by Nephron-Sparing Surgery or Cytoreductive Nephrectomy in Locally Advanced and Metastatic Renal Cell Carcinomas
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was closed due to extremely low accrual, as well as a change in care when using the study drug.
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-2961
Record Dates: First submitted 2017-06-12; First posted 2017-06-16 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Renal Cell Carcinoma; Metastatic Kidney Cancer
Keywords: Kidney Cancer; Immunotherapy; Renal Cell Carcinoma; Cryoablation; Metastatic Renal Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — pembrolizumab; Cryosurgery; Nephrectomy

STUDY DESIGN:
Intervention Model Description: This is a longitudinal single armed open-label trial for advanced (stage II and above with multiple tumors or vena cava) and metastatic Renal Cell Carcinoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): Advanced (stage II and above with multiple tumors or vena cava) and metastatic Renal Cell Carcinoma will be first treated with cryoablation on a large primary tumor and then given 200 mg pembrolizumab every 3-week for 3 cycles, followed by cytoreductive or partial/radical nephrectomy. After the surgery, patients will resume pembrolizumab for additional 5 cycles or up to a total of 2 years if a partial response is observed at the discretion of the treating medical oncologist or urologist until a complete tumor remission, disease progression, unacceptable toxicity, subject refusal, or subject death due to any cause.
  Interventions: Drug: Pembrolizumab Injection [Keytruda]; Procedure: Cryoablation; Procedure: Nephrectomy

INTERVENTIONS:
Drug: Pembrolizumab Injection [Keytruda] — Same as arm description
  Other Names: Pembrolizumab
Procedure: Cryoablation — Cryoablation uses liquid argon in metal needles to freeze tumors. Tumor cells are ruptured due to the forming ice crystals and die. Cryoablation is standardly used in tumors less then 4cm in diameter.
Procedure: Nephrectomy — Nephrectomy is the surgical excision of either the entire kidney or a small portion of the kidney. Nephrectomy is standardly used to treat renal cell cancer.
  Other Names: Partial Nephrectomy; Radical Nephrectomy; Nephron Sparring Surgery

SUMMARY:
Patients will undergo a screening process as per standard of care to identify disease type and severity. Careful history and physical examination will also take place to rule out major heart, lung, or kidney disease and pregnancy that may affect how they will respond to the treatment. Patients with advanced (stage II and above with multiple tumors or tumors within vessels) and metastatic Renal Cell Carcinoma will be first treated with cryoablation on a large primary tumor and then given 200 mg pembrolizumab every 3-weeks 3 cycles , followed by partial/radical nephrectomy. Pembrolizumab is a biologic drug that adheres to the cell death receptors on white blood cells preventing there death and leading to an increased immunologic response. Cryoablation will be used in these patients to initially trigger and immune response to cancerous cells that is then magnified by the drug. After the surgery, patients will resume pembrolizumab for additional 5 cycles or up to a total of 2 years if a partial response is observed at the discretion of the treating medical oncologist or urologist until complete tumor remission, disease progression, unacceptable toxicity, patient refusal, or patient death due to any cause.

DETAILED DESCRIPTION:
Baseline procedures:

Each patient will undergo a careful history and physical examination to rule out major cardiac, pulmonary or renal disease. All subjects will undergo:

1. Baseline biopsy of a secondary tumor or a metastatic tumor at the time of cryoablation. Tumor specimens will also be collected during surgery (cytoreductive, partial or total nephrectomy).
2. One or more optional biopsies at day 53, day 106 and day 169 after cryoablation.
3. Blood samples: will be collected at baseline before or at time of cryoablation, at the end of the second cycle of pembrolizumab treatment and during surgery (cytoreductive, partial or total nephrectomy) for evaluation of biomarkers and pharmacokinetic analyses.
4. Complete radiologic assessment in the form of CT scan at baseline and a CT scan after the third cycle of pembrolizumab followed by routine imaging every 6 weeks as is consistent with the standard of care for mRCC. 5. Routine laboratory analysis: basic metabolic panel (BMP), liver function panel (LFTs) and complete blood count (CBC), will be collected prior to each cycle of pembrolizumab administration and at the time of cryoablation and cytoreductive or partial/total nephrectomy.

Cryoablation:

Patients will be asked to have nothing by mouth during at least 8 hours prior to ablation. Patients will only be taken for cryoablation if INR is <1.5, PTT is within normal limits and platelet count is greater than 50,000/microL. Preoperative imaging, namely contrast enhanced CT scan, will be used to assess the tumor proximity to local structures. Number of cryoprobes utilized will be determined by the size, geometry, and morphology of the primary tumor. CT guidance will be used to place the cryoprobes 1 to 1.5 cm apart.

Two 10 minute freeze cycles with an intervening 8 minute thawing period will be used in accordance with data indicating improved efficacy with the double-freeze thaw cycle. The size of the iceball created will be consistent with a tumor-free margin of at least 5-10 mm. CT scans at 3-4 minute intervals will be used to assure adequate margins.

Pembrolizumab:

Pembrolizumab treatment will begin 1 day following cryoablative treatment and will continue until a complete tumor remission, disease progression, unacceptable toxicity, subject refusal, or subject death due to any cause.

Surgery After 3 cycles (9 weeks) of pembrolizumab therapy, patients will undergo partial/ radical or cytoreductive nephrectomy of the primary renal tumor.

Duration of follow-up Subjects will be followed for a total of 24 months. Subjects removed from treatment due to unacceptable adverse events will be followed until resolution or stabilization of adverse event. Follow up will be every 8 weeks (+2 weeks) from study registration with imaging studies and physical exam every 8 weeks for the first 8 months, then every 12 weeks (+ 2 weeks) until 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be >18 years of age on day of signing informed consent.
3. Have measurable disease based on RECIST 1.1.
4. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.
5. Have a performance status of 0 or 1 on the ECOG Performance Scale.
6. Demonstrate adequate organ function as defined in days of treatment initiation.
7. All screening labs should be performed within 10 days of treatment initiation.
8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female subjects of childbearing potential (Section 5.7.2) must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 120 days after the last dose of study medication.

   Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
10. Male subjects of childbearing potential (Section 5.7.1) must agree to use an adequate method of contraception as outlined in Section 5.7.1- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has known history of, or any evidence of active, non-infectious pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
15. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
17. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
18. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | 24 weeks after cryoablation
  Tumor responses to pembrolizumab and cryoablation combination followed by partial, radical or cytoreductive nephrectomy on secondary lesions. The tumor responses will be defined by CT images according to RECIST version 1.1., and reviewed by an experienced oncologist. The primary endpoint will be percentage of patients who achieve a best ORR, including both partial and complete responses.

SECONDARY OUTCOMES:
Progression-free Survival | Follow-up will be for 24 months
  PFS is defined as time from cryoablation initiation to time of first documented disease progression or death due to any cause.
Overall Survival | Follow-up will be for 24 months
  OS is time from cryoablation to death due to any cause. OS will be assessed at standard clinic visits.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Landman, MD, Principal Investigator — UC Irvie Department of Urology
Locations (1):
- UC Irvine Health Department of Urology, Orange, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] Hruby GW, Fine JK, Landman J. Ultrasound-guided percutaneous ablation of a renal mass in a renal allograft. Urology. 2006 Oct;68(4):891.e5-6. doi: 10.1016/j.urology.2006.05.019. PMID 17070386
- [Background] Ames CD, Vanlangendonck R, Venkatesh R, Gonzales FC, Quayle S, Yan Y, Humphrey PA, Landman J. Enhanced renal parenchymal cryoablation with novel 17-gauge cryoprobes. Urology. 2004 Jul;64(1):173-5. doi: 10.1016/j.urology.2004.02.033. PMID 15245965
- [Background] Okhunov Z, Juncal S, Ordon M, George AK, Lusch A, del Junco M, Nguyentat M, Lobko II, Kavoussi L, Landman J. Comparison of outcomes in patients undergoing percutaneous renal cryoablation with sedation vs general anesthesia. Urology. 2015 Jan;85(1):130-4. doi: 10.1016/j.urology.2014.09.013. Epub 2014 Nov 14. PMID 25440762
- [Background] Lusch A, Graversen JA, Liss MA, Landman J. Ablative techniques: Radiofrequency and cryotherapy, which is the best? Arch Esp Urol. 2013 Jan-Feb;66(1):71-8. PMID 23406802
- [Background] Waitz R, Solomon SB, Petre EN, Trumble AE, Fasso M, Norton L, Allison JP. Potent induction of tumor immunity by combining tumor cryoablation with anti-CTLA-4 therapy. Cancer Res. 2012 Jan 15;72(2):430-9. doi: 10.1158/0008-5472.CAN-11-1782. Epub 2011 Nov 22. PMID 22108823
- [Background] Zeng Z, Shi F, Zhou L, Zhang MN, Chen Y, Chang XJ, Lu YY, Bai WL, Qu JH, Wang CP, Wang H, Lou M, Wang FS, Lv JY, Yang YP. Upregulation of circulating PD-L1/PD-1 is associated with poor post-cryoablation prognosis in patients with HBV-related hepatocellular carcinoma. PLoS One. 2011;6(9):e23621. doi: 10.1371/journal.pone.0023621. Epub 2011 Sep 1. PMID 21912640
- [Background] Hamid O, Robert C, Daud A, Hodi FS, Hwu WJ, Kefford R, Wolchok JD, Hersey P, Joseph RW, Weber JS, Dronca R, Gangadhar TC, Patnaik A, Zarour H, Joshua AM, Gergich K, Elassaiss-Schaap J, Algazi A, Mateus C, Boasberg P, Tumeh PC, Chmielowski B, Ebbinghaus SW, Li XN, Kang SP, Ribas A. Safety and tumor responses with lambrolizumab (anti-PD-1) in melanoma. N Engl J Med. 2013 Jul 11;369(2):134-44. doi: 10.1056/NEJMoa1305133. Epub 2013 Jun 2. PMID 23724846
- [Background] Massari F, Santoni M, Ciccarese C, Santini D, Alfieri S, Martignoni G, Brunelli M, Piva F, Berardi R, Montironi R, Porta C, Cascinu S, Tortora G. PD-1 blockade therapy in renal cell carcinoma: current studies and future promises. Cancer Treat Rev. 2015 Feb;41(2):114-21. doi: 10.1016/j.ctrv.2014.12.013. Epub 2015 Jan 6. PMID 25586601
- [Background] Zeelenberg IS, van Maren WW, Boissonnas A, Van Hout-Kuijer MA, Den Brok MH, Wagenaars JA, van der Schaaf A, Jansen EJ, Amigorena S, Thery C, Figdor CG, Adema GJ. Antigen localization controls T cell-mediated tumor immunity. J Immunol. 2011 Aug 1;187(3):1281-8. doi: 10.4049/jimmunol.1003905. Epub 2011 Jun 24. PMID 21705625
- [Background] Keerthikumar S, Gangoda L, Liem M, Fonseka P, Atukorala I, Ozcitti C, Mechler A, Adda CG, Ang CS, Mathivanan S. Proteogenomic analysis reveals exosomes are more oncogenic than ectosomes. Oncotarget. 2015 Jun 20;6(17):15375-96. doi: 10.18632/oncotarget.3801. PMID 25944692